CLINICAL TRIAL: NCT01538303
Title: Microvascular Dysfunction in AMI and Its Relation to Outcome
Brief Title: Microvascular Dysfunction in Acute Myocardial Infarction (AMI) and Its Relation to Outcome
Status: Completed | Type: Observational
Sponsor: Catharina Ziekenhuis Eindhoven (Other)
Responsible Party: Principal Investigator, Inge Wijnbergen, MD, Catharina Ziekenhuis Eindhoven
Other Study IDs: NL-3793806011
Record Dates: First submitted 2012-02-20; First posted 2012-02-24 (Estimated); Last update posted 2023-02-10 (Actual); Status verified 2023-02

CONDITIONS: ST Segment Elevation Myocardial Infarction
Keywords: STEMI; absolute flow; microvascular resistance
MeSH Terms: conditions — ST Elevation Myocardial Infarction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- measurement absolute flow and resistance

SUMMARY:
The purpose of this study is first to evaluate absolute myocardial blood flow and resistance over time in the acute and sub-acute phase of myocardial infarction and second, to correlate these parameters to preservation of left ventricular function and long-term outcome.

DETAILED DESCRIPTION:
In acute myocardial infarction, early restoration of epicardial and myocardial blood flow is of paramount importance to limit infarct size and create optimum conditions for favorable long-term outcome.

Presently, restoration of epicardial blood flow is preferably obtained by primary percutaneous coronary intervention (PPCI). PPCI is the treatment of choice for patients with acute myocardial infarction who can be admitted sufficiently fast to a hospital equipped for this type for treatment.

Successful restoration of epicardial blood flow by PPCI is possible in approximately 90% of all patients. Nevertheless, in a number of these patients myocardial hypoperfusion persists due to moderate or severe microvascular dysfunction.

The terminology "no reflow" is often used for this condition. Microvascular thromboembolism, spasm, or intramyocardial oedema are suggested to be responsible for this condition and probably all of these three phenomena play a role. Besides that, inflammatory response of the myocardium can be involved with neutrophil plugging of the capillaries, further compromising restoration of normal myocardial blood flow and function.

It is well known that in patients in whom myocardial reperfusion is absent or limited, despite adequate epicardial reperfusion, prognosis is poor and more severe left ventricular dysfunction can be expected in comparison to those patients in whom also microvascular reperfusion after PPCI is restored. Therefore, it is beyond doubt that knowledge about the actual state of the microvasculature and myocardial (re)perfusion shortly after PPCI, is important from a prognostic point of view.

Moreover, if microvascular reperfusion is still limited immediately after myocardial infarction, but recovers quickly in the days thereafter, this might have important implications for long-term prognosis.

Lastly, knowledge about microvascular reperfusion in the acute phase can be important with respect to choice of adjunct mechanical or medical therapy, such as intra aortic balloon pumping (IABP), Gp IIb/IIIa inhibitors or continuation of nitroglycerine.

Despite this undisputed importance of microvascular perfusion and function in the acute phase of myocardial infarction, its assessment has been difficult so far and has been hampered by a number of methodological and technical shortcomings.It should be realized in this context that the function of the microvasculature in general (and specifically in acute myocardial infarction) can be characterized by myocardial blood flow and resistance.

Recently, the investigators have developed a new technique for measuring absolute coronary and myocardial blood flow and absolute and relative coronary and myocardial resistance This has paved the way to study microvascular function in acute myocardial infarction immediately after epicardial reperfusion by PPCI and in the days thereafter.

ELIGIBILITY:
Inclusion Criteria:

* STEMI < 12 hours
* > 10mm ST-segment deviation
* culprit lesion in proximal or mid segment of a coronary artery with a reference diameter > 3.0mm by visual estimation.
* hemodynamically stable.

Exclusion Criteria:

* Age > 75 years
* cardiogenic shock or pre-shock
* Patients in whom no access to the coronary circulation can be obtained by the femoral artery or in whom femoral access was problematic.
* Patients with previous myocardial infarction in the culprit area of with previous bypass surgery
* Tortuous coronary arteries or complex or long-lasting primary PCI
* Severe concomitant disease or conditions with a life expectancy of less than one year
* Inability to understand and give informed consent either in first instance on the table or in second instance on the coronary care unit.
* Other known myocardial diseases, such as moderate or severe left ventricular hypertrophy or cardiomyopathy
* Pregnancy

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population consists of patients with STEMI either in our own hospital either referred by other hospitals or the ambulance.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2012-03 (Actual); Primary Completion 2012-10 (Actual); Study Completion 2012-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nico Pijls, MD, PhD, Principal Investigator — Catharina Ziekenhuis Eindhoven
Locations (1):
- Catharina Hospital Eindhoven, Eindhoven, North Brabant, Netherlands